CLINICAL TRIAL: NCT01079325
Title: A Phase 2b Repeat Dosing Clinical Trial of SB-509 in Subjects With Moderately Severe Diabetic Neuropathy
Brief Title: Clinical Trial of SB-509 in Subjects With Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB-509-0901
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Polyneuropathy
Keywords: Diabetic neuropathy; Diabetes Type 1 or 2; Moderately severe sensorimotor diabetic polyneuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Neuropathies | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB-509 (Experimental)
  Interventions: Drug: SB-509
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: SB-509 — SB-509 60 mg, 3 treatments, and 5 months treatment period
  Arms: SB-509
Other: Saline
  Other Names: 30 ml saline, 3 treatments
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the clinical effects of the investigational drug, SB-509, in subjects with diabetic neuropathy.

DETAILED DESCRIPTION:
SB-509 contains the gene (DNA-a kind of biological "blueprint") for a protein. When a researcher injects SB-509 into your legs, the drug enters the muscle and nerve cells around the injection site and causes these cells to make a protein. This protein causes your cells to increase production of another protein called vascular endothelial growth factor (VEGF), which may improve the structure and function of nerves. In addition, there are changes in the levels of additional proteins in your cells. These proteins function to promote the growth of cells, are structures in cells, help synthesize products, and affect immune cells, and some have unknown functions. This increase in your own VEGF proteins may protect and repair the damaged nerves caused by diabetic neuropathy.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of Diabetes Mellitus Type I or II for at least 12 months
* Clinical signs and symptoms of moderate to severe diabetic sensory-motor polyneuropathy of the lower extremities for at least 6 months that are not otherwise attributed to an etiology other than diabetes
* Measurable sural and peroneal response bilaterally
* HgbA1C level ≤ 10%
* LDL cholesterol ≤ 160 mg/dL
* Blood pressure ≤ 140/90 mm Hg
* Body mass index (BMI) ≤ 38

Key Exclusion Criteria:

* Moderate to severe ischemic heart disease or any history of congestive heart failure, or have had a myocardial infarction within the previous 6 months
* Evidence of cardiac enlargement and/or congestive heart failure
* Current diabetic foot or leg ulcer, gangrene in the lower extremity, or any amputation of the lower extremity
* History of malignancy, except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for at least 5 years
* Immune or immunodeficiency disorders or expected to require immunosuppressants for 30 days prior to, during, and for 30 days following administration of the investigational drug product
* History of or current proliferative retinopathy, macular edema or retinal neovascularization
* Pre-cancerous conditions or benign tumors which have the potential for clinically significant growth due to VEGF stimulation
* Family history of inherited neuropathy (e.g. Charcot Marie Tooth, Hereditary Predisposition to Pressure Palsy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2009-11; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To compare the effect of SB-509 versus placebo in subjects with moderately severe diabetic neuropathy (DN) on sural Nerve Conduction Velocity (NCV) at six-months | 6 months

SECONDARY OUTCOMES:
To evaluate the effect of SB-509 on Neuropathy Impairment Score - Lower Limb (NIS-LL), motor Nerve Conduction Velocity (NCV), Quantitative Sensory Testing (QST), Intraepidermal Nerve Fiber Density (IENFD), and Lower Extremity Neurological Sensory Exam | 12 months
To evaluate the effect of SB-509 using a multi-endpoint analysis that includes NIS-LL, Sural NCV, and IENFD | 12 months
To evaluate the safety of SB-509 in subjects with moderately severe diabetic neuropathy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Winson Tang, MD, Study Director — Sangamo BioSciences, Inc
Locations (31):
- United States (31):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Chino, California
  - Fresno, California
  - La Jolla, California
  - Los Angeles, California
  - National City, California
  - San Francisco, California
  - Walnut Creek, California
  - Boulder, Colorado
  - DeLand, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Winston-Salem, North Carolina
  - Tulsa, Oklahoma
  - Greer, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.sangamo.com